CLINICAL TRIAL: NCT01448096
Title: Multi-center Phase II Study of the Combination of R-CHOP (RItuximab Plus Cyclophosphamide, Adriamycin, Vincristine, and Prednisolone) and Prophylactic Intrathecal Chemotherapy With Methotrexate in Patients With CD20+ Primary Breast Diffuse Large B-cell Lymphoma
Brief Title: Study in Patients With Primary Breast Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: Consortium for Improving Survival of Lymphoma (Other)
Responsible Party: Principal Investigator, Ho-Young Yhim, Principal investigator, Chonbuk National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chonbuk058
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Large B Cell Diffuse Lymphoma
Keywords: primary breast diffuse large B cell lymphoma; rituximab; prophylactic intrathecal chemotherapy; CNS recurrence
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- primary breast DLBCL (Experimental): isolated breast involvement with or without nodal disease
  Interventions: Drug: Rituximab; Procedure: Prophylactic intrathecal chemotherapy

INTERVENTIONS:
Drug: Rituximab — R-CHOP21 consist of rituximab (375 mg/m2), cyclophosphamide (750 mg/m2), doxorubicin (50 mg/m2), and vincristine (1.4 mg/m2, a maximum of 2mg), administered intravenously on day 1 and 100 mg oral prednisone on days 1 through 5.
Procedure: Prophylactic intrathecal chemotherapy — Prophylactic intrathecal chemotherapy using methotrexate (12mg total dose) will be performed

SUMMARY:
The purpose of this study is to clarify the impact of rituximab on clinical outcomes in patients with primary breast diffuse large B-cell lymphoma and also to investigate the role of prophylactic intrathecal chemotherapy using methotrexate for reducing central nervous system (CNS) recurrence.

DETAILED DESCRIPTION:
Primary breast diffuse large B-cell lymphoma (DLBCL) is a rare presentation of non-Hodgkin's lymphoma. A significant risk of contralateral breast involvement and a tendency for central nervous system (CNS) progression have been identified in previous studies. Optimal treatment strategies for primary breast DLBCL have remained undefined, although the combination of anthracycline-based chemotherapy and radiotherapy may be considered to be the best treatment option in these studies. However, despite the administration of aggressive treatment, prognosis is still poor, even in localized disease, with 5-year progression-free survival rates of approximately 50% to 65% in most series. Therefore, other therapeutic options must be explored.

During the last decade, several studies have shown that rituximab plus CHOP or CHOP-like chemotherapy significantly improves clinical outcomes of patients with DLBCL. However, the relevance of rituximab in the management of this rare extranodal lymphoma has never been studied. Moreover, several studies have also suggested the possibility that prophylactic intrathecal chemotherapy might be effective in reducing CNS recurrence.

Thus, this trial is designed to prospectively evaluate the treatment strategy, which addressed the safety and efficacy of a combined therapy that included R-CHOP21 and prophylactic intrathecal chemotherapy using methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20 positive primary breast DLBCL
* age ≤ 70
* No prior chemotherapy or radiotherapy for DLBCL
* Performance status (ECOG) ≤ 2
* Cardiac ejection fraction ≥ 50 % as measured by MUGA or 2D ECHO without clinically significant abnormalities
* Adequate renal function: serum creatinine level < 2 mg/dL (177 μmol/L)
* Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value, Bilirubin < 2 X upper normal value
* Adequate BM functions: hemoglobin ≥ 9 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL
* A negative serum or urine pregnancy test prior to treatment must be available both for pre menopausal women and for women who are < 1 years after the onset of menopause
* Life expectancy more than 6 months
* Informed consent

Exclusion Criteria:

* other subtype primary breast non-Hodgkin's lymphoma than DLBCL
* secondary breast DLBCL
* Patients with a known history of HIV seropositivity or HCV (+). Patients who have HBV (+) are eligible. However, primary prophylaxis using antiviral agents (i.e. lamivudine) is recommended for HBV carrier to prevent HBV reactivation during whole treatment period.
* Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions

  * Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
  * History of significant neurologic or psychiatric disorders including dementia or seizures
  * Active uncontrolled infection (viral, bacterial or fungal infection)
  * Other serious medical illnesses
* Known hypersensitivity to any of the study drugs or its ingredients (i.e., hypersensitivity to Polysorbate 20, CHO cell products, or recombinant human antibodies)
* Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-08; Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
progression-free survival | From the date of treatment until the date of disease progression or death from any cause (minimum 2 years)

SECONDARY OUTCOMES:
overall survival | From the date of treatment until the date of death from any cause (minimum 2 years)
Number of patients with CNS recurrence | From the date of treatment until the date of CNS recurrrence (minimum 2 years)
Number of patients with adverse events | From the first date of treatment until 30 days after the last treatment
  safety of a combined treatment of R-CHOP21 and prophylactic intrathecal chemotherapy according to the NCI-CTCAE ver.3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Kwak, MD, PhD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

REFERENCES:
- [Background] Yhim HY, Kim JS, Kang HJ, Kim SJ, Kim WS, Choi CW, Eom HS, Kim JA, Lee JH, Won JH, Shim H, Huh J, Lee DH, Suh C, Kwak JY. Matched-pair analysis comparing the outcomes of primary breast and nodal diffuse large B-cell lymphoma in patients treated with rituximab plus chemotherapy. Int J Cancer. 2012 Jul 1;131(1):235-43. doi: 10.1002/ijc.26352. Epub 2011 Aug 30. PMID 21823120
- [Background] Yhim HY, Kang HJ, Choi YH, Kim SJ, Kim WS, Chae YS, Kim JS, Choi CW, Oh SY, Eom HS, Kim JA, Lee JH, Won JH, Shim H, Lee JJ, Sung HJ, Kim HJ, Lee DH, Suh C, Kwak JY. Clinical outcomes and prognostic factors in patients with breast diffuse large B cell lymphoma; Consortium for Improving Survival of Lymphoma (CISL) study. BMC Cancer. 2010 Jun 22;10:321. doi: 10.1186/1471-2407-10-321. PMID 20569446